CLINICAL TRIAL: NCT00030966
Title: A Randomized, Double-Blind, Placebo-Controlled, Parallel-Group, Multicenter Study to Determine the Safety and Efficacy of Natalizumab, When Added to Avonex® (Interferon Beta-1a), in Subjects With Relapsing-Remitting Multiple Sclerosis
Brief Title: Safety and Efficacy of Natalizumab in Combination With Avonex in the Treatment of Multiple Sclerosis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Biogen (Industry)
Collaborators: Elan Pharmaceuticals (Industry)
Responsible Party: Biogen Idec MD, Biogen Idec
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: C-1802
Record Dates: First submitted 2002-02-15; First posted 2002-02-18 (Estimated); Last update posted 2009-06-18 (Estimated); Status verified 2009-06

CONDITIONS: Multiple Sclerosis, Relapsing-Remitting
Keywords: Multiple Sclerosis; MS
MeSH Terms: conditions — Multiple Sclerosis, Relapsing-Remitting; Multiple Sclerosis | interventions — Natalizumab

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Group 1 (Experimental): Adding natalizumab monthly infusion to Avonex weekly injection for up to 116 weeks.
  Interventions: Drug: Natalizumab
- Group 2 (Placebo Comparator): Adding placebo monthly infusion to Avonex weekly injection for up to 116 weeks.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Natalizumab — Natalizumab, 300 mg, monthly IV infusion for up to 116 weeks.
  Other Names: Tysabri
  Arms: Group 1
Drug: Placebo — Placebo monthly infusion for up to 116 weeks.
  Arms: Group 2

SUMMARY:
The purpose of this study is to determine if natalizumab in combination with AVONEX is safe and effective in delaying progression of individuals diagnosed with relapsing remitting Multiple Sclerosis (MS).

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of MS as defined by McDonald et al, criteria, # 1- 4
* Between the ages of 18 and 55, inclusive
* Baseline EDSS score between 0.0 and 5.0, inclusive
* Have been treated with Avonex for at least the 12 months prior to randomization
* Have experienced at least one relapse (while on Avonex) within the 12 months prior to randomization.
* Cranial MRI scan demonstrating lesions consistent with MS.
* Have given written informed consent to participate in the study.

Exclusion Criteria:

* Primary progressive, secondary progressive, or progressive relapsing MS.
* MS relapse has occurred within 50 days of randomization
* A clinically significant infectious illness within 30 days prior to randomization
* History of, or abnormal lab result, indicative of significant disease, that in the opinion of the investigator, would preclude the administration of a recombinant humanized antibody immunomodulating agent or Avonex for 116 weeks.
* History of severe allergic or anaphylactic reactions or known drug hypersensitivity.
* Unable to perform the Timed 25-Foot Walk, 9HPT and PASAT 3
* Abnormal blood tests at Screening Visit

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 1200 (Actual)
Dates: Start 2002-01; Primary Completion 2005-04 (Actual); Study Completion 2005-12 (Actual)

PRIMARY OUTCOMES:
Primary objectives of this study are to determine if natalizumab is effective in reducing the rate of clinical relapse at 1 year and in slowing the progression of disability at 2 years as measured by EDSS. | 1 year and 2 years

SECONDARY OUTCOMES:
If this combination reduces MRI lesions and the overall rate of clinical relapses | 1 year and 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Michael Panzara, MD, MPH, Study Director — Biogen; Richard A Rudick, MD, Principal Investigator — The Cleveland Clinic
Locations (88):
- United States (72):
  - University of Alabama-Birmingham, Department of Neurology, Birmingham, Alabama
  - Phoenix Neurological Associates, Ltd., Phoenix, Arizona
  - University of Arkansas For Medical Sciences, Little Rock, Arkansas
  - University of California - Irvine, Irvine, California
  - USC MS Comprehensive Care Center, Los Angeles, California
  - Kaiser-Permanente Medical Center, Redwood City, California
  - MS Center at UCSF, San Francisco, California
  - Healthsouth Rehabilitation Hospital, Colorado Springs, Colorado
  - University of Colorado MS Center, Denver, Colorado
  - Griffin Hospital, Derby, Connecticut
  - Georgetown Univesity Hospital, Research Pharmacy, Washington D.C., District of Columbia
  - George Washington University MS Center, Washington D.C., District of Columbia
  - North Ridge NeuroScience Center, Fort Lauderdale, Florida
  - Maitland Neurology, Maitland, Florida
  - University of Miami, Department of Neurology, Miami, Florida
  - The Multiple Sclerosis Center of Atlanta, Atlanta, Georgia
  - Marietta Neurological Associates, Marietta, Georgia
  - Northwestern University, Department of Neurology, Chicago, Illinois
  - Rush-Presbyterian St. Luke's Medical Center, Chicago, Illinois
  - Alexian Brothers Center for Clinical Research, Elk Grove Village, Illinois
  - Loyola Medical Center, Maywood, Illinois
  - Consultants in Neurology Northbrook, Northbrook, Illinois
  - Springfield Clinic Neuroscience Institute, Springfield, Illinois
  - Indiana University Medical Center, Indianapolis, Indiana
  - Mercy Hospital Outpatient Pharmacy, Des Moines, Iowa
  - LSU Neurolgoy Clinic in New Orleans, New Orleans, Louisiana
  - Maine Neurology, Scarborough, Maine
  - University of Maryland Hospital, Department of Neurology, Baltimore, Maryland
  - Brigham and Women's Hospital, Boston, Massachusetts
  - University of Massachusetts Memorial Medical Center, Worcester, Massachusetts
  - Henry Ford Hospital, Detroit, Michigan
  - Michigan State University MS Clinic, East Lansing, Michigan
  - Michigan Institute for Neurological Disorders, Farmington Hills, Michigan
  - Noran Neurological Clinic, Minneapolis, Minnesota
  - University of Mississippi Medical Center, Jackson, Mississippi
  - St. John's Mercy Medical Center, St Louis, Missouri
  - Bernard W. Gimbel MS Center, Teaneck, New Jersey
  - Upstate Clinical Research, LLC, Albany, New York
  - Albany Medical Center, Albany, New York
  - Maimonides Medical Center, Division of Neurology, Brooklyn, New York
  - Buffalo General Hospital, Department of Neurology, Buffalo, New York
  - MS Care Center, New York, New York
  - St. Luke's Roosevelt Hospital, MS Research & Treatment Center, New York, New York
  - New York Hospital - Cornell Medical Center, New York, New York
  - New York State Psychiatric Institution, New York, New York
  - Strong Health Pharmacy Services, Rochester, New York
  - Staten Island University Hospital, Staten Island, New York
  - University Hospital at Stony Brook, Stony Brook, New York
  - SUNY Upstate Medical University, Syracuse, New York
  - MS Center at Carolinas Medical Center, Charlotte, North Carolina
  - Raleigh Neurology Associates, Raleigh, North Carolina
  - Wake Forest University School of Medicine, Department of Neurology, Winston-Salem, North Carolina
  - Riverhills Neurology, Cincinnati, Ohio
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Providence Saint Vincent Medical Center, Portland, Oregon
  - Geisinger Medical Center, Danville, Pennsylvania
  - Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania
  - Greenstein Neurology Associates & MS Institute, Philadelphia, Pennsylvania
  - Allegheny Singer Research Institute, Pittsburgh, Pennsylvania
  - University of Pittsburgh, Department of Neurology, Pittsburgh, Pennsylvania
  - University of Tennessee - Memphis, Memphis, Tennessee
  - Vanderbilt Medical Center, Nashville, Tennessee
  - Option Care Infusion, Dallas, Texas
  - UTSW Medical School, Dallas, Texas
  - Baylor Methodist International MS Center, Houston, Texas
  - Central Texas Neurology, Round Rock, Texas
  - Fletcher Allen Health Care, Burlington, Vermont
  - University of Virginia Health Sciences, Charlottesville, Virginia
  - Neurological Associates, Inc., Richmond, Virginia
  - Virginia Mason Medical Center, Seattle, Washington
  - MS Research Center, Seattle, Washington
  - St. Francis Hospital, Center for Neurological Disorders, Milwaukee, Wisconsin
- Austria (2):
  - Universitatsklinik fur Neurologie, Graz
  - Universitatsklinik fur Neurologie, Innsbruck
- Belgium (2):
  - Hopital Universitaire U.L.B. Erasme, Brussels
  - Elisabeth Ziekenhuis, Sijsele
- France (2):
  - Hopital Pellegrin Tripode, Neurologie, Bordeaux
  - Hopital neurologique Pierre Werth, Lyon
- Germany (7):
  - Judisches Krankenhaus, Berlin
  - Universitaetsklinikum Giessen, Oberarzt Neurologie, Giessen
  - Medizinische Hochschule Hannover, Neurologische Klinik, Hanover
  - Neurologische Abteilung, Henningsdorf
  - Städtische Kliniken Osnabrück, Osnabrück
  - Asklepios Klinik Schildautal, Seesen/Harz
  - Fachbereich Neurologie und Klinische Neurophysiologie, Wiesbaden
- Israel (2):
  - Hadassah Hebrew Uni Hospital, Department of Neurology, Jerusalem
  - Sheba Medical Center, MS Center, Tel Litwinsky
- Universita di Genova, Clinica Neurologica, Genova, Italy

REFERENCES:
- [Result] Rudick RA, Stuart WH, Calabresi PA, Confavreux C, Galetta SL, Radue EW, Lublin FD, Weinstock-Guttman B, Wynn DR, Lynn F, Panzara MA, Sandrock AW; SENTINEL Investigators. Natalizumab plus interferon beta-1a for relapsing multiple sclerosis. N Engl J Med. 2006 Mar 2;354(9):911-23. doi: 10.1056/NEJMoa044396. PMID 16510745
- [Derived] Strijbis EM, Coerver E, Mostert J, van Kempen ZLE, Killestein J, Comtois J, Repovic P, Bowen JD, Cutter G, Koch M. Association of age and inflammatory disease activity in the pivotal natalizumab clinical trials in relapsing-remitting multiple sclerosis. J Neurol Neurosurg Psychiatry. 2023 Oct;94(10):792-799. doi: 10.1136/jnnp-2022-330887. Epub 2023 May 12. PMID 37173129
- See also: The web site of the National Multiple Sclerosis Society, an organization dedicated to providing information to individuals with MS, their families and healthcare providers. — http://www.nationalmssociety.org
- See also: MSActiveSource.com is a resource for news, information and disease management for all individuals touched by multiple sclerosis. This site is sponsored by Biogen. — http://www.msactivesource.com